CLINICAL TRIAL: NCT03872921
Title: Double-blind, Randomized, Placebo-controlled, Phase III Study Comparing norUrsodeoxycholic Acid Capsules With Placebo in the Treatment of Primary Sclerosing Cholangitis
Brief Title: norUrsodeoxycholic Acid vs Placebo in PSC
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NUC-5/PSC
Record Dates: First submitted 2019-03-08; First posted 2019-03-13 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — 24-norursodeoxycholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- norUrsodeoxycholic acid (Experimental): norUrsodeoxycholic acid 250mg capsules, 6 capsules/day for 2 years
  Interventions: Drug: norUrsodeoxycholic Acid
- Placebo to norUrsodeoxycholic acid (Placebo Comparator): norUrsodeoxycholic acid 250mg Placebo-capsules, 6 capsules/day for 2 years
  Interventions: Drug: norUrsodeoxycholic Acid

INTERVENTIONS:
Drug: norUrsodeoxycholic Acid — oral treatment
  Other Names: NUC

SUMMARY:
Double-blind, randomized, multi-center, placebo-controlled, comparative, phase III trial. The study will be conducted with two treatment groups in the form of a parallel group comparison and will serve to compare oral treatment with either 1500 mg/d norursodeoxycholic acid capsules or placebo capsules for the treatment of Primary Sclerosing Cholangitis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* verified PSC
* Liver Biopsy available for Review
* If pre-treated with UDCA Patient must be on stable dose not exceeding 20mg/kg/bw
* Patients with or without concomittant IBD

Exclusion Criteria:

* History or presence of other concomitant liver diseases
* Presence of Cholangiocarcinoma
* Secondary causes of Sclerosing Cholangitis
* Small Duct Cholangitis in the absence of large duct disease
* Any known relevant infectious disease
* Abnormal renal function
* Any active malignant disease
* Known intolerance/hypersensitivity to study drug

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
superiority of norursodeoxycholic acid (norUDCA) compared to placebo in the treatment of Primary Sclerosing Cholangitis (PSC) | 2 years
  prevention of disease progression assessed by partial normalization of serum Alkaline Phosphatase (s-ALP) levels in patients with PSC
Show superiority of norursodeoxycholic acid (norUDCA) compared to placebo in the treatment of Primary Sclerosing Cholangitis (PSC) | 2 years
  prevention of disease progression assessed by liver histology

CONTACTS AND LOCATIONS:
Overall Officials: Michael Trauner, MD, Principal Investigator — Medical University of Vienna, Department of Internal Medicine III
Locations (2):
- Medical University of Vienna, Department of Internal Medicine III, Vienna, Austria
- Medical School Hannover, Hanover, Lower Saxonia, Germany

IPD SHARING:
Plan to Share IPD: No
It is not yet decided which data will be made available. Neither a time Frame can be indicated yet.